CLINICAL TRIAL: NCT05864183
Title: Screening for Risk Factors of Prediabetes Among Adults Patients at Sohag University Hospital
Brief Title: Screening for Risk Factors of Prediabetes Among Adult Patients at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nermin Fathy Ezzat, internal medicine resident at faculty of medicine Sohag university, Sohag University
Other Study IDs: Soh-Med-23-04-20MS
Record Dates: First submitted 2023-04-19; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Urinalysis; Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: prediabetic
  Interventions: Diagnostic Test: HbA1c; Diagnostic Test: lipid profile; Diagnostic Test: CBC; Diagnostic Test: Alb/cr ratio; Diagnostic Test: serum creatinine .; Diagnostic Test: CRP; Diagnostic Test: urine analysis; Diagnostic Test: ECG; Diagnostic Test: fundus examination
- control group: non prediabetic
  Interventions: Diagnostic Test: HbA1c; Diagnostic Test: lipid profile; Diagnostic Test: CBC; Diagnostic Test: Alb/cr ratio; Diagnostic Test: serum creatinine .; Diagnostic Test: CRP; Diagnostic Test: urine analysis; Diagnostic Test: ECG; Diagnostic Test: fundus examination

INTERVENTIONS:
Diagnostic Test: HbA1c — HbA1c will be measured for all patients to minimize the risk of developing diabetes or its complications .
Diagnostic Test: lipid profile — lipid profile will be measured for all patients to minimize the risk of developing diabetes or its complications .
Diagnostic Test: CBC — CBC will be measured for all patients to minimize the risk of developing diabetes or its complications
Diagnostic Test: Alb/cr ratio — Alb/cr will be measured for all patients to minimize the risk of developing diabetes or its complications
Diagnostic Test: serum creatinine . — serum creatinine will be measured for all patients to minimize the risk of developing diabetes or its complications
Diagnostic Test: CRP — CRP will be measured for all patients to minimize the risk of developing diabetes or its complications
Diagnostic Test: urine analysis — urine analysis will be measured for all patients to minimize the risk of developing diabetes or its complications
Diagnostic Test: ECG — ECG will be done for all patients to minimize the risk of developing diabetes or its complications
Diagnostic Test: fundus examination — fundus examination will be done for all patients to minimize the risk of developing diabetes or its complications

SUMMARY:
* Prediabetes is an intermediate state of hyperglycemia with glycemic parameters above normal but below the diabetes threshold..
* during the average 3 years of follow-up Prediabetes is diagnosed based on laboratory tests: fasting plasma glucose level (100-125 mg/dl) ;HbA1c, (5.7-6.4%) or plasma glucose level after an oral glucose tolerance test ( 140-199 mg/dl).
* Reports estimate that more than 470 million people will have prediabetes by 2030.
* According to an expert panel of the American Diabetes Association, up to 70% of individuals with prediabetes will eventually develop diabetes.
* Observational evidence suggests as association between prediabetes and complications of diabetes such early nephropathy(10%) , small fiber neuropathy(18-25 %), early retinopathy (8-12%) and risk of macrovascular disease (52%) .
* Screening for prediabetes is designed to save lives or enhance an individual's quality of life by early detection so that screening will minimize the risk of developing diabetes or its complications .

DETAILED DESCRIPTION:
* In this case control study we aim to screen for risk factors of prediabetes among adult patients to minimize the risk of developing diabetes or its complications .
* Prediabetes screening is also required to minimize medical costs such as hospitalization, outpatient care, surgery, medications, and laboratory test costs .
* Several studies had shown efficacy of lifestyle interventions in diabetes prevention by targeting obesity with increase in physical activity and dietary changes with a relative risk reduction of 40%-70% in adults with prediabetes ,also there is increasing evidence to prove the efficacy of pharmacotherapy in prevention of diabetes in adults with prediabetes

ELIGIBILITY:
Inclusion Criteria:

* Adult patient above 18 years old .

Exclusion Criteria:

* all patients known to be diabetics .
* pregnancy .
* chronic depleting diseases,
* Those who were taking drugs known to influence blood glucose levels e.g. metformin, thiazolidinedione and steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted to Sohag University hospital at period of admission 18 years or older wihe exclusion of patients known to be diabetics , pregnants , chronic depleting diseases patients , those who were taking drugs known to influence blood glucose levels e.g. metformin, thiazolidinedione and steroids.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
comparison between the measurement of HbA1c in normal non prediabetics and prediabetics at Sohag university hospital . | 6 months
  analysis of HbA1c measurements and compare the results in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tabak AG, Herder C, Rathmann W, Brunner EJ, Kivimaki M. Prediabetes: a high-risk state for diabetes development. Lancet. 2012 Jun 16;379(9833):2279-90. doi: 10.1016/S0140-6736(12)60283-9. Epub 2012 Jun 9. PMID 22683128
- [Background] Beulens J, Rutters F, Ryden L, Schnell O, Mellbin L, Hart HE, Vos RC. Risk and management of pre-diabetes. Eur J Prev Cardiol. 2019 Dec;26(2_suppl):47-54. doi: 10.1177/2047487319880041. PMID 31766914
- [Result] Vas PRJ, Alberti KG, Edmonds ME. Prediabetes: moving away from a glucocentric definition. Lancet Diabetes Endocrinol. 2017 Nov;5(11):848-849. doi: 10.1016/S2213-8587(17)30234-6. Epub 2017 Aug 3. No abstract available. PMID 28781065